CLINICAL TRIAL: NCT03452631
Title: Spontaneous Haematomas of Psoas Occurring in Intensive Care: Incidence, Patient Characteristics and Treatment, a Retrospective Study
Brief Title: Spontaneous Haematomas of Psoas Occurring in Intensive Care
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6838
Record Dates: First submitted 2018-02-26; First posted 2018-03-02 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Psoas Hematomas
Keywords: Psoas hematomas

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Psoas hematomas are a rare and potentially lethal pathology whose incidence in resuscitation is unknown. The pathophysiology of this pathology is not known to date.

ELIGIBILITY:
Inclusion Criteria:

* Major patients
* Psoas hematoma diagnosed during hospitalization

Exclusion Criteria:

* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with psoas hematoma diagnosed during hospitalization
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Number of psoas hematomas | 72 hours after admission to intensive care

CONTACTS AND LOCATIONS:
Overall Officials: Julie HELMS, MD, Study Director — University Hospital, Strasbourg, France
Locations (1):
- Service de Réanimation médicale, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No